CLINICAL TRIAL: NCT02910609
Title: International Experience in Timing And Choices of Treatment For Ductal Closure in Patent Ductus Arteriosus: INTERPDA Trial
Brief Title: International Experience in Timing And Choices for Ductal Closure in Patent Ductus Arteriosus:INTERPDA Trial
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Omer Erdeve, Ankara University, Clinical Profesor, Ankara University
Other Study IDs: Ankara University
Record Dates: First submitted 2016-09-12; First posted 2016-09-22 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Patent Ductus Arteriosus
Keywords: preterm; patent ductus arterioles; treatment
MeSH Terms: conditions — Ductus Arteriosus, Patent; Premature Birth | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Management at PN 3-7 days: Preterm infants with hemodynamically significant PDA confirmed by echocardiography and are treated at 3-7 days of their life
  Interventions: Device: Echocardiography
- Management after PN 7 days: Preterm infants with hemodynamically significant PDA confirmed by echocardiography and are treated beyond 7 days of their life
  Interventions: Device: Echocardiography

INTERVENTIONS:
Device: Echocardiography — Echocardiography is a kind of ultrasound test that shows the inner structure and functions of the heart in both groups.

SUMMARY:
The three options for the treatment of patent ductus arterioles (PDA) in preterm infants are conservative approach, pharmacological intervention and surgical ligation. There is not any randomized-controlled trial that demonstrates the superiority of these approaches in preterm infants.

DETAILED DESCRIPTION:
Patent ductus arteriosus (PDA), of which incidence is inversely related to gestational age and birth weight, is one of the the most common conditions among preterm infants.

In recent years, the use of antenatal steroids, postnatal surfactant, noninvasive ventilation strategies and low oxygen saturation targets have affected the incidence of hemodynamically significant PDA (HSPDA). There is not any consensus about the best approach on the clinical management of PDA in preterm infants. Over past years, the management of HSPDA shifted to aggressive medical and surgical intervention from conservative treatment, but conservative treatment approach has been mainly concerned again nowadays.

Today, the three options for the treatment of PDA in preterm infants are conservative approach, pharmacological intervention and surgical ligation. There is not any randomized-controlled trial that demonstrates the superiority of these approaches in preterm infants. Many countries including developed countries only give recommendations, instead of publishing guidelines, on screening, timing of treatment and treatment choices of PDA, because of the differences on management of PDA between the centers even within a single center.

Timing of PDA treatment and treatment choices at preterm infants born before 28 gestation weeks' differ in our country also in many countries over the world. In this study, it is aimed to record the managements of PDA detected beyond postnatal 3 days, to compare the effects of the managements at postnatal 3-7 days and after 7 days on closure, surgical ligation rates and side effects of drugs.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at 24 0/7-28 6/7 gestation weeks'
* PDA detected with ductal diameter equal or greater than 1.5 mm and LA/Ao equal or greater than 1.5 on echocardiography at or after postnatal 72 hours of life

Exclusion Criteria:

* Infants died before 72 hours of life
* Infants detected PDA but treated before 72 hours of life

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants born at 24 0/7-28 6/7 gestation weeks' who were performed echocardiography at or after postnatal 72 hours of life, and detected ductal diameter equal or greater than 1.5 mm and LA/Ao equal or greater than 1.5 are the candidates for the study. The management of PDA and the other data of these infants will be registered to online registry system.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Spontan closure rate | 3 months
  Rate of patients with spontaneous ductal closure

SECONDARY OUTCOMES:
Surgical ligation rate | 3 months
  rate of patients who need surgical ligation for hemodynamically significant ductus
Complications of prematurity | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ömer Erdeve, Professor, Principal Investigator — Ankara University

IPD SHARING:
Plan to Share IPD: No
No data individual data will be shared